CLINICAL TRIAL: NCT05307172
Title: Precision Medicine Approach to Unravel the Risk Factors for Renal, Cardiovascular, Ophthalmologic, Neurologic and Hepatic Complications of Metabolic Disorders
Acronym: PRECIMETAB
Status: Withdrawn | Type: Observational
Why Stopped: No inclusion within 2 years of approval by CPP
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Hospitalier Universitaire, Amiens (Other); Biobanque de Picardie (Unknown)
Responsible Party: Sponsor
Other Study IDs: C21-13; 2021-A02192-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2021-12

CONDITIONS: Chronic Kidney Diseases; Diabetes; Obesity
Keywords: Chronic Kidney Diseases; Diabetes; Precision Medicine; Biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The study requires the collection of blood, urine, and a hair strand for analyses specifically dedicated to the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There is currently no way to predict the progression of chronic kidney disease in patients with metabolic disease(s). Furthermore, the mechanisms responsible for the development and/or progression of complications remain largely unknown.

In order to identify the predictive factors and/or mechanisms involved in the different complications of these diseases, we propose an approach coupling :

* a classical phenotypic characterization (clinical, biological, imaging) of the patients
* high-throughput screening of the genome, transcriptome, metabolome, proteome, and immunophenotyping.

According to our hypothesis, this approach should allow :

* Early detection of complications
* Classification of patients in homogeneous groups of patients with identical evolution
* Identification of the molecular mechanisms involved.

DETAILED DESCRIPTION:
Eligible patients will be detected during one of their consultations at the precision medicine center of the Amiens-Picardy University Hospital. They will be informed of the proposed research pathway during a care consultation. After a period of reflection, patients who accept this pathway will be included and a written consent form will be collected.

The inclusion visit will be scheduled at the precision medicine center of the Amiens-Picardy University Hospital and will take place during a day hospital (HDJ) which is part of a routine care pathway (neurological, cardiovascular, hepatic and renal primary prevention). At the time of inclusion, the informed consent will be signed by the investigator as well as by the patient The collection of data obtained during the patient's routine care will be performed by a physician from the Precision Medicine Center and a clinical research nurse and will be recorded in the patient's medical record.

Biological samples for the research (additional blood volume, urine) will be taken in conjunction with those for the routine check-up.

A hair strand of approximately 100 hairs (approx. 2 mm diameter) will be collected at the inclusion visit. This sample will be optional and will be subject to a specific authorization from the patient on the consent form.

Biological samples intended for research will be sent by the department's staff to the Biobank of Picardie (CHU Amiens-Picardie) for processing and storage.

The follow-up of the patient will be done strictly within the framework of his care adapted to his pathology. No visits will be made specifically for research purposes. The schedule of follow-up visits for the study corresponds to the visits usually scheduled as part of patient care: at 1 year after the inclusion visit (A1), at 4 years (A4) and at 7 years (A7).

In summary: One year after the inclusion visit, the patient will have a clinical and biological evaluation including a measurement of renal function to determine the rate of decline of glomerular filtration rate in order to classify the patient as a non-progressor, a moderate-progressor, or a rapid-progressor (see primary endpoints). The rate of decline of GFR will be correlated with clinical, biological, genetic and environmental data collected at patient inclusion, by means of dedicated questionnaires, biological results collected and analyses performed on research samples taken during the patient inclusion visit. The prognostic power of the classic clinical and biological criteria and of the new biomarkers discovered during the study to predict the patient's all-cause evolutionary profile will be evaluated́ by hazard ratio and 95% confidence interval. This reassessment will then be repeated at each visit until the end of the study.

Follow-up visits will be conducted in the same manner as the inclusion visit. The collection of data obtained during the routine care follow-up will be performed by a Precision Medicine Center physician and a clinical research nurse and will be recorded in the patient's medical record.

Additional biological samples (additional volume of blood, urine) will be taken during the care samples to meet the research objectives.

The occurrence of a pregnancy during the follow-up period will not constitute an exclusion criterion. The patient will be able to continue her participation in the study.

Failure to complete one of the follow-up visits will not be considered an early exit from the research. The patient will be scheduled for the next protocol visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons, male or female, age ≥ 18 and ≤ 65 years
* Persons able to understand the information provided and to object to it (at the discretion of the investigator)
* Patient affiliated to a social security system.
* Patient willing to sign an informed consent form
* Patient with the following metabolic profile Diabetic (of any type) treated or not (diabetes will be defined by a fasting blood glucose > 7mM or a HbA1c > 6.5% or by the use of an antidiabetic treatment) AND/OR Obese patient (BMI > 30 kg/m2) treated or not
* Patient with evidence of renal parenchymal damage defined by an albuminuria/creatinuria ratio ≥ 3 mg/mmol (30mg/g), AND/OR a glomerular filtration rate estimated by the CKD-EPI (eDFG) formula classifying the patient as stage 2 to 3a of the KDIGO classification (i.e., 90ml/min/1.73 m2 > GFR > 45ml/min), AND/OR a renal lithiasis

Exclusion Criteria:

* Patient deprived of liberty
* Person subject to a legal protection measure (guardianship, curatorship or safeguard of justice)
* Patient refusing to participate in the study
* Pregnant, parturient or nursing woman
* Patient in emergency situation
* Patient with advanced chronic kidney disease defined as GFR < 45ml/min/1.73 m².
* Contraindication to Iohexol injection
* Patient with or who has had any of the following complications: symptomatic coronary artery disease, symptomatic peripheral arterial disease, previous stroke, previous myocardial infarction, heart failure ≥ stage B, dementia, liver fibrosis, hepatocarcinoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, suffering from obesity and/or diabetes and presenting signs of renal parenchymal suffering, referred to the Amiens-Picardie University Hospital for monitoring of the renal function and screening in primary prevention of associated neurological, hepatic and cardiovascular comorbidities.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-03 (Estimated); Primary Completion 2032-05-03 (Estimated); Study Completion 2032-05-03 (Estimated)

PRIMARY OUTCOMES:
the rate of annual decline in glomerular filtration rate (GFR year n+1 - GFR year n) measured by iohexol clearance | from day 1 of inclusion, up to 7 years
  The rate of annual decline in glomerular filtration rate (GFR year n+1 - GFR year n) measured by iohexol clearance, which will distinguish three groups of patients:
  * Those with physiological (age-related) annual decline: <2ml/min per 1.73 m²/year (non-progressors),
  * Those with moderate annual decline ≥2 and <5 ml/min per 1.73 m²/year (moderate progressors)
  * Those with rapid annual decline ≥5 ml/min per 1.73 m²/year (rapid progressors)

SECONDARY OUTCOMES:
The evolution of vascular status | from day 1 of inclusion, up to 7 years
  The evolution of vascular status will be assessed by blood pressure (SBP, DBP, DBP), central pressure and vascular stiffnes
Major cardiovascular event | from day 1 of inclusion, up to 7 years
  Major cardiovascular event defined as cardiovascular death, myocardial infarction, hospitalization for heart failure, stroke (ischemic or hemorrhagic), or acute limb ischemia
microvascular event | from day 1 of inclusion, up to 7 years
  -A microvascular event defined as the occurrence of complicated peripheral sensory neuropathy and/or the occurrence of proliferative retinopathy or metabolic blindness
Cognitive performance | from day 1 of inclusion, up to 7 years
  Cognitive performance will be assessed by neuropsychological testing. A decline in cognitive performance will be defined as a decrease of at least 1.5 standard deviations on at least 1 neuropsychological test within a cognitive domain from the neuropsychological assessment performed at inclusion
The onset of dementia defined as a cognitive disorder | from day 1 of inclusion, up to 7 years
  - The onset of dementia defined as a cognitive disorder as evidenced by the neuropsychological assessment performed at the end of the study resulting in a loss of functional autonomy in activities of daily living as measured by a loss of at least one point on the ADL scale (DSMV).deviations on at least 1 neuropsychological test within a cognitive domain from the neuropsychological assessment performed at inclusion
The occurrence of severe liver damage | from day 1 of inclusion, up to 7 years
  The occurrence of severe liver damage will be defined by :
  fibrosis, cirrhosis, hepatocarcinoma, or death of hepatic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'AMIENS - Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No